CLINICAL TRIAL: NCT06840769
Title: A Phase I, Open Label, Single Dose, Two Parts Study in Male and Female Healthy Subjects to Assess the Safety and Pharmacokinetics of Fosnetupitant 235 mg Administered as IV Bolus and of Derived Netupitant and Netupitant Metabolites
Brief Title: A Clinical Trial to Assess Safety and Pharmacokinetics of Fosnetupitant 235 mg and Metabolites in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: PNET-22-08
Record Dates: First submitted 2025-02-11; First posted 2025-02-21 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteers
Keywords: Helsinn; PNET-22-08; Fosnetupitant; Netupitant
MeSH Terms: interventions — Solutions; netupitant, palosentron drug combination

STUDY DESIGN:
Intervention Model Description: Open label, single dose, two parts (part A and part B), safety and pharmacokinetic phase I study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Study Part A - cohort 1 (Experimental): Fosnetupitant free base 235 mg administered as single 30 min intravenous infusion or 235 mg fosnetupitant/0.25 mg palonosetron in 20 mL injection solution administered undiluted as a single 30 min intravenous infusion
  Interventions: Drug: Fosnetupitant 235 mg solution; Drug: Akynzeo solution
- Study Part A - cohort 2 (Experimental): Fosnetupitant free base 235 mg administered as single 15 min intravenous infusion
  Interventions: Drug: Fosnetupitant 235 mg solution
- Study Part A - cohort 3 (Experimental): Fosnetupitant free base 235 mg administered as single 5 min intravenous infusion
  Interventions: Drug: Fosnetupitant 235 mg solution
- Study Part A - cohort 4 (Experimental): Fosnetupitant free base 235 mg administered as single 2 min intravenous infusion
  Interventions: Drug: Fosnetupitant 235 mg solution

INTERVENTIONS:
Drug: Fosnetupitant 235 mg solution — Fosnetupitant free base 235 mg (corresponding to 260 mg of the chloride hydrochloride salt) in 20 mL ready to use injectable solution for intravenous administration
  Other Names: Helsinn Fosnetupitant solution
Drug: Akynzeo solution — 235 mg fosnetupitant (corresponding to 260 mg of the chloride hydrochloride salt) / 0.25 mg palonosetron in 20 mL injectable solution
  Other Names: IV Akynzeo®
  Arms: Study Part A - cohort 1

SUMMARY:
This clinical trial will include two parts, i.e., Part A and Part B.

The goal of the Part A is to define the shortest safe and tolerable duration of an intravenous injection of Fosnetupitant 235 mg solution among 4 durations tested in male and female adult healthy volunteers. In study part A, researchers will compare Fosnetupitant 235 mg solution to Akynzeo® solution.

The duration determined in Part A will be investigated in study Part B.

The Part B of the study was not performed.

DETAILED DESCRIPTION:
The registered product Akynzeo® (235 mg fosnetupitant/0.25 mg palonosetron) solution for intravenous injection, used before chemotherapy, is to be diluted up to a final volume of 50 mL and administered during 30 min infusion. With the aim to facilitate and improve the use of this kind of products, the Sponsor Helsinn focused on the development of a ready to use solution, not requiring additional dilutions, and to be administered as a bolus injection. The product developed by Helsinn is a liquid formulation for infusion, containing exclusively fosnetupitant 235 mg free base.

Aim of the present open label, single dose, two parts (part A and part B) phase I study is to evaluate the safety and the pharmacokinetic profile of this new product, i.e., Fosnetupitant 235 mg ready to use solution for intravenous injection. In addition, the pharmacokinetic profile of fosnetupitant, netupitant (fosnetupitant is rapidly converted in netupitant after intravenous administration) and netupitant metabolites (M1, M2 and M3) will be investigated after a 30-min infusion of the registered Akynzeo® liquid formulation.

Part A of the study:

In cohort 1, 10 healthy volunteers will receive a dose of Fosnetupitant 235 mg solution as a one single 30-min intravenous infusion and additional 10 subjects will receive a single intravenous dose of Akynzeo® solution as a one single 30-min intravenous infusion, according to a parallel group design.

In each of 3 consecutive cohorts (cohorts 2, 3 and 4), 10 healthy volunteers will receive a single intravenous dose of Fosnetupitant 235 mg solution at a predefined infusion duration and will be sequentially treated as 3 subgroups of 3, 3, and 4 subjects, respectively.

A staggered approach with decreasing infusion time duration will be applied, from cohort 1 to cohort 4, to the administration of Fosnetupitant free base 235 mg solution, as follows:

Cohort 1: 30 min Cohort 2: 15 min Cohort 3: 5 min Cohort 4: 2 min

At the end of cohort 1 and of each subgroup of cohorts 2, 3 and 4, safety and tolerability results will be evaluated by the Investigator and the study Sponsor Medical Expert. Predefined stopping rules will be considered for deciding about continuing with the next cohort treatment and a shorter injection duration of Fosnetupitant 235 mg solution. Specifically, after cohort 1, if the injection duration of 30 min proves to be safe and well tolerated, 15 min injection duration will be tested in cohort 2. If the injection duration of 15 min proves to be safe and well-tolerated, 5 min injection duration will be tested in cohort 3. If the injection duration of 5 min proves to be safe and well tolerated, a 2 min injection will be tested in cohort 4.

The selected shortest (safe and tolerable) injection duration determined in Part A will be investigated in study Part B.

The study was prematurely terminated after the end of Part A and study Part B was not performed.

ELIGIBILITY:
Inclusion criteria

1. Informed consent: signed written informed consent before inclusion in the study
2. Sex and Age: healthy men/women volunteers, 18-55 years old (inclusive)
3. Body Mass Index (BMI): 18.5-30 kg/m2 inclusive
4. Vital signs: systolic blood pressure 100-139 mmHg, diastolic blood pressure 50-89 mmHg, pulse rate 50-99 bpm, measured after 5 min at rest in the sitting position
5. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study
6. Contraception and fertility (women only): women of childbearing potential defined as a non-menopausal woman who has not had a bilateral oophorectomy or medically documented ovarian failure and/or at risk for pregnancy must agree, signing the informed consent form, to use a highly effective method of contraception throughout the study and to continue for 14 days after the last dose of the study treatment. Highly effective contraceptive measures include:

   1. Hormonal oral, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit.
   2. A non-hormonal intrauterine device [IUD] for at least 2 months before the screening visit
   3. A sterile or vasectomized sexual partner
   4. True (long-term) heterosexual abstinence, defined as refraining from heterosexual intercourse when this is in line with the preferred and usual lifestyle of the subject, while periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), lactational amenorrhea and withdrawal are not acceptable.

   Women of non-child-bearing potential or in post-menopausal status defined as such when there is either:
   1. 12 months of spontaneous amenorrhea or
   2. 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL or
   3. 6 weeks documented postsurgical bilateral oophorectomy with or without hysterectomy will be admitted. For all women, pregnancy test result must be negative at screening and admission (Day -1).
7. Contraception (men only): men will either be sterile or agree to use one of the following approved methods of contraception from the first study drug administration until at least 14 days after the last administration, also in case their partner is currently pregnant:

   1. A male condom with spermicide
   2. A sterile sexual partner or a partner in post-menopausal status for at least one year
   3. Use by the female sexual partner of an IUD, a female condom with spermicide, a contraceptive sponge with spermicide, a diaphragm with spermicide, a cervical cap with spermicide, or hormonal oral, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit Men must accept to inform their partners of the participation in the clinical study. Furthermore, they will not donate sperm from the date of the informed consent form's signature, throughout the study, and for at least 14 days after the last dose of the study treatment. These requirements are based upon the availability and results of reproductive toxicity data.

Exclusion criteria

1. 12-leads Electrocardiogram (ECG) (supine position): clinically significant abnormalities at screening. With regards to QTc, the following will be considered as exclusion criterion: mean corrected QT (QTcF) > 450 ms. HR < 50 or > 99 bpm. PR < 100 or >220 ms. QRS > 120 ms. Relevantly abnormal T-wave patterns
2. Physical examination findings: clinically significant abnormal physical findings which could interfere with the objectives of the study
3. Laboratory analyses: clinically significant abnormal laboratory values at screening, indicative of physical illness or suggesting the subject's exclusion, in his/her best interest
4. Allergy: ascertained or presumptive hypersensitivity to the active principle and/or formulations' ingredients; history of anaphylaxis to drugs or allergic reactions in general, which the investigator considers may affect the outcome of the study
5. Diseases: significant history, in the opinion of the Investigator, of renal, hepatic, gastrointestinal, cardiovascular (in particular, heart failure, hypokalemia, family history of Long QT Syndrome, history of superficial thrombophlebitis or deep vein thrombosis), respiratory, skin, hematological, endocrine or neurological diseases that may interfere with the aim of the study
6. Medications: medications, including over the counter (OTC) medications and herbal remedies in the 2 weeks before the first visit of the study. Hormonal contraceptives for women are allowed
7. CYP3A4 inducers and inhibitors: use of any inducer or inhibitor of CYP3A4 enzymes (drugs, food, herbal remedies) in the 28 days or in the 7 days, respectively, before the planned first study drug administration and during the whole study
8. Investigative drug studies: participation in the evaluation of any investigational product for 3 months before this study. The 3-month interval is calculated as the time between the first calendar day of the month that follows the last visit of the previous study and the first day of the present study
9. Blood donation or significant blood loss: blood donations or significant blood loss in the 3 months before the first visit of this study
10. Drug, alcohol, caffeine, tobacco: history of drug, alcohol [>1 drink/day for women and >2 drinks/day for men, defined according to the USDA Dietary Guidelines 2020-2025 (11)], caffeine (>5 cups coffee/tea/day) or tobacco abuse (≥10 cigarettes/day)
11. Drug test: positive result at the urine drug screening test at screening or Day -1
12. Alcohol test: positive salivary alcohol test at Day -1
13. Diet: abnormal diets (<1600 or >3500 kcal/day) or substantial changes in eating habits in the 4 weeks before screening; vegetarians
14. Pregnancy (women only): positive or missing pregnancy test at screening or Day -1, pregnant or lactating women
15. Netupitant studies: enrolment in a previous study of netupitant or fosnetupitant (alone or in combination with palonosetron)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-06-17 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milko Radicioni, Principal Investigator — Cross Research S.A.
Locations (1):
- CROSS Research S.A., Arzo, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: No
No need to share IPD

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the Phase I Unit from 12 June 2023 to 14 October 2023 and enrolled in the study from 17 June 2023 to 16 October 2023.
Pre-assignment Details: Fifty (50) subjects were included in the study and received the treatment as planned.
Groups:
- Study Part A - Cohort 1 - Akynzeo: 10 subjects were included in the study as planned and received the injection of Akynzeo solution in 30 min.
- Study Part A - Cohort 1 - Fosnetupitant: 10 subjects were included in the study as planned and received the injection of Fosnetupitant 235 mg solution in 30 min.
- Study Part A - Cohort 2: 10 subjects were included in the study as planned and received the injection of Fosnetupitant 235 mg solution in 15 min.
- Study Part A - Cohort 3: 10 subjects were included in the study as planned and received the injection of Fosnetupitant 235 mg solution in 5 min.
- Study Part A - Cohort 4: 10 subjects were included in the study as planned and received the injection of Fosnetupitant 235 mg solution in 2 min.
Period: Overall Study
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Started | 10 | 10 | 10 | 10 | 10
Completed | 9 | 10 | 10 | 10 | 10
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4 | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (8.9) | 40.7 (8.2) | 38.9 (13.2) | 37.9 (10.8) | 38.1 (13.5) | 37.5 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 3 | 3 | 4 | 20
  Male | 6 | 4 | 7 | 7 | 6 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 1
  White | 10 | 10 | 9 | 8 | 9 | 46
  More than one race | 0 | 0 | 0 | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Switzerland | 10 | 10 | 10 | 10 | 10 | 10
Body weight [Mean (Standard Deviation); unit: kilograms] | 65.94 (9.50) | 69.83 (15.15) | 71.98 (13.16) | 75.20 (11.24) | 71.30 (11.66) | 70.85 (12.16)
Height [Mean (Standard Deviation); unit: centimeters] | 171.0 (8.1) | 168.0 (9.3) | 170.1 (8.4) | 174.0 (10.4) | 169.4 (9.1) | 170.5 (9.0)
Body mass index [Mean (Standard Deviation); unit: kilograms/square meters] | 22.46 (2.20) | 24.49 (3.36) | 24.69 (2.65) | 24.74 (2.26) | 24.83 (3.42) | 24.24 (2.86)

OUTCOME MEASURES:

1. Primary Outcome: Study Part A: Number of Treatment-emergent Adverse Events
Description: Number of treatment-emergent adverse events (TEAEs) collected up to 24 h post-dose.
Time Frame: From screening visit (day of informed consent signature) up to 24 h after the investigational medicinal product administration (a maximum of 21 days)
Measure: Number; unit: Number of TEAE
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Number of TEAE | 7 | 4 | 3 | 1 | 4

2. Primary Outcome: Study Part A: Number of Subjects With Treatment-emergent Adverse Events
Description: Number of subjects with treatment-emergent adverse events (TEAEs) collected up to 24 h post-dose.
Time Frame: as for outcome 1
Measure: Number; unit: Number of subjects with TEAE
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Number of subjects with TEAE | 5 | 3 | 2 | 1 | 4

3. Primary Outcome: Study Part A: Type of Treatment-emergent Adverse Events
Description: Type of treatment-emergent adverse events (TEAEs) collected up to 24 h post-dose.
Time Frame: as for outcome 1
Measure: Number; unit: Number of TEAE
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Number of TEAE
  Gastrointestinal disorders | 2 | 1 | 0 | 0 | 0
  General disorders and administration site conditions | 2 | 2 | 0 | 1 | 0
  Nervous system disorders | 2 | 1 | 2 | 0 | 4
  Psychiatric disorders | 1 | 0 | 0 | 0 | 0
  Investigations | 0 | 0 | 1 | 0 | 0

4. Secondary Outcome: Study Part A: Systolic Blood Pressure
Description: Systolic blood pressure in mmHg measured after 5 min at rest in sitting position
Time Frame: Screening visit/day -1 (enrolment day)/day 1 (treatment day) at pre-administration, at the end of administration and 1, 2, 4, 24 h after the end of administration/final visit (7 days after the treatment)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
mmHg
  Screening visit | 119.7 (9.4) | 118.8 (9.7) | 122.6 (12.5) | 122.6 (12.5) | 119.1 (8.9)
  Day -1 (enrolment day) | 113.1 (6.2) | 116.7 (6.6) | 122.0 (12.5) | 122.0 (12.5) | 118.8 (9.7)
  Day 1 (treatment day) at pre-administration | 112.5 (8.2) | 112.8 (12.9) | 114.2 (12.2) | 114.2 (12.2) | 115.6 (10.7)
  Day 1 (treatment day) at the end of administration | 107.7 (12.3) | 111.5 (8.5) | 113.6 (10.6) | 113.6 (10.6) | 113.2 (13.5)
  Day 1 (treatment day) at 1 h after the end of administration | 110.4 (8.2) | 111.7 (10.6) | 113.4 (11.9) | 113.4 (11.9) | 112.3 (10.2)
  Day 1 (treatment day) at 2 h after the end of administration | 106.6 (6.9) | 109.8 (11.6) | 114.1 (10.8) | 114.1 (10.8) | 112.4 (7.6)
  Day 1 (treatment day) at 4 h after the end of administration | 108.3 (10.5) | 107.6 (9.5) | 113.8 (12.7) | 113.8 (12.7) | 109.8 (9.6)
  Day 1 (treatment day) at 24 h after the end of administration | 108.5 (8.2) | 112.9 (11.7) | 116.7 (10.8) | 116.7 (10.8) | 115.8 (10.6)
  Final visit (7 days after the treatment) | 114.4 (9.3) | 111.1 (11.8) | 116.2 (8.7) | 116.2 (8.7) | 120.5 (10.9)

5. Secondary Outcome: Study Part A: Diastolic Blood Pressure
Description: Diastolic blood pressure in mmHg measured after 5 min at rest in sitting position
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
mmHg
  Screening visit | 72.3 (6.5) | 76.8 (6.9) | 80.4 (8.0) | 80.4 (8.0) | 76.7 (7.5)
  Day -1 (enrolment day) | 68.9 (8.6) | 77.7 (5.8) | 76.1 (7.0) | 76.1 (7.0) | 74.8 (6.9)
  Day 1 (treatment day) at pre-administration | 72.1 (9.0) | 74.9 (9.2) | 76.0 (10.1) | 76.0 (10.1) | 71.9 (10.5)
  Day 1 (treatment day) at the end of administration | 62.4 (11.1) | 71.7 (8.3) | 75.2 (10.1) | 75.2 (10.1) | 70.1 (9.3)
  Day 1 (treatment day) at 1 h after the end of administration | 63.9 (6.4) | 73.4 (8.3) | 76.7 (8.8) | 76.7 (8.8) | 72.5 (7.2)
  Day 1 (treatment day) at 2 h after the end of administration | 64.5 (8.5) | 72.8 (7.3) | 74.8 (11.2) | 74.8 (11.2) | 71.5 (9.2)
  Day 1 (treatment day) at 4 h after the end of administration | 65.9 (6.6) | 68.9 (8.8) | 76.6 (9.8) | 76.6 (9.8) | 70.7 (8.5)
  Day 1 (treatment day) at 24 h after the end of administration | 67.0 (9.4) | 72.7 (7.9) | 77.5 (8.8) | 77.5 (8.8) | 73.2 (7.7)
  Final visit (7 days after the treatment) | 70.1 (7.2) | 74.4 (7.5) | 77.7 (7.1) | 77.7 (7.1) | 77.4 (6.4)

6. Secondary Outcome: Study Part A: Pulse Rate
Description: Pulse rate in bpm measured after 5 min at rest in sitting position
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: Beats/min
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Beats/min
  Screening visit | 60.9 (7.3) | 65.3 (7.8) | 61.0 (10.5) | 61.0 (10.5) | 68.3 (7.3)
  Day -1 (enrolment day) | 68.4 (8.9) | 74.9 (8.6) | 75.6 (11.7) | 75.6 (11.7) | 77.7 (8.8)
  Day 1 (treatment day) at pre-administration | 60.0 (5.6) | 62.4 (8.6) | 59.0 (9.4) | 59.0 (9.4) | 65.2 (7.2)
  Day 1 (treatment day) at the end of administration | 58.3 (7.5) | 64.2 (8.6) | 59.5 (7.7) | 59.5 (7.7) | 62.0 (10.1)
  Day 1 (treatment day) at 1 h after the end of administration | 59.3 (10.4) | 62.8 (5.4) | 59.3 (7.8) | 59.3 (7.8) | 62.4 (8.9)
  Day 1 (treatment day) at 2 h after the end of administration | 56.4 (6.8) | 61.4 (6.8) | 58.5 (7.8) | 58.5 (7.8) | 62.1 (9.2)
  Day 1 (treatment day) at 4 h after the end of administration | 56.8 (7.2) | 62.7 (7.5) | 56.4 (7.2) | 56.4 (7.2) | 62.8 (7.9)
  Day 1 (treatment day) at 24 h after the end of administration | 58.8 (9.8) | 65.5 (7.9) | 60.9 (9.0) | 60.9 (9.0) | 67.8 (6.5)
  Final visit (7 days after the treatment) | 56.8 (8.1) | 62.9 (6.8) | 61.5 (7.4) | 61.5 (7.4) | 72.3 (10.5)

7. Secondary Outcome: Study Part A: Weight
Description: Body weight in kilograms
Time Frame: Screening visit (day of informed consent signature)/final visit (7 days after the treatment)
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Kilograms
  Screening visit | 65.94 (9.50) | 69.83 (15.15) | 71.98 (13.16) | 71.98 (13.16) | 71.30 (11.66)
  Final visit (7 days after the treatment) | 66.68 (9.49) | 70.08 (14.67) | 72.44 (13.72) | 72.44 (13.72) | 71.40 (11.48)

8. Secondary Outcome: Study Part A: Full Physical Examination Through Apparatus/Systems Check
Description: General appearance, Chest/respiratory, Gastrointestinal, Head, eyes, ears, nose and throat, Heart/cardiovascular, Lymph nodes, Metabolic/endocrine, Musculoskeletal/extremities, Neck (including thyroid), Neurological/psychiatric, Skin/dermatologic systems are checked. Any abnormalities are recorded.
Time Frame: Screening visit (day of informed consent signature)/final visit (7 days after the treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  Screening visit: Normal | 10 | 7 | 9 | 10 | 9
  Screening visit: Abnormal not clinically significant | 0 | 3 | 1 | 0 | 1
  Final visit (7 days after the treatment): Normal | 10 | 7 | 10 | 10 | 10
  Final visit (7 days after the treatment): Abnormal not clinically significant | 0 | 3 | 0 | 0 | 0

9. Secondary Outcome: Study Part A: Short Physical Examination Through Apparatus/Systems Check
Description: General appearance, Chest/respiratory, Heart/cardiovascular, Lymph nodes, Neurologic/psychiatric, Skin/dermatologic systems are checked. Any abnormalities are recorded.
Time Frame: Day 2 (24 h after the end of investigational product administration)
Measure: Count of Participants; unit: Participants
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  Normal | 9 | 7 | 10 | 10 | 10
  Abnormal not clinically significant | 1 | 3 | 0 | 0 | 0

10. Secondary Outcome: Study Part A: ECGs - Heart Rate
Description: Heart rate in beats/min recorded in supine position after 5 min at rest
Time Frame: Screening visit/ day 1 (treatment day) at pre-administration, at the end of administration and 1, 2, 4, 24 h after the end of administration/final visit (7 days after the treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  Screening visit: Normal | 3 | 4 | 2 | 3 | 5
  Screening visit: Abnormal not clinically significant | 7 | 6 | 8 | 7 | 5
  Day 1 (treatment day) at pre-administration: Normal | 1 | 4 | 2 | 2 | 2
  Day 1 (treatment day) at pre-administration: Abnormal not clinically significant | 9 | 6 | 8 | 8 | 8
  Day 1 (treatment day) at the end of administration: Normal | 2 | 3 | 2 | 2 | 2
  Day 1 (treatment day) at the end of administration: Abnormal not clinically significant | 8 | 7 | 8 | 8 | 8
  Day 1 (treatment day) at 1 h after the end of administration: Normal | 1 | 2 | 2 | 1 | 2
  Day 1 (treatment day) at 1 h after the end of administration: Abnormal not clinically significant | 9 | 8 | 8 | 9 | 8
  Day 1 (treatment day) at 2 h after the end of administration: Normal | 0 | 2 | 2 | 2 | 2
  Day 1 (treatment day) at 2 h after the end of administration: Abnormal not clinically significant | 10 | 8 | 8 | 8 | 8
  Day 1 (treatment day) at 4 h after the end of administration: Normal | 1 | 2 | 1 | 1 | 2
  Day 1 (treatment day) at 4 h after the end of administration: Abnormal not clinically significant | 9 | 8 | 9 | 9 | 8
  Day 1 (treatment day) at 24 h after the end of administration: Normal | 0 | 4 | 2 | 3 | 5
  Day 1 (treatment day) at 24 h after the end of administration: Abnormal not clinically significant | 10 | 6 | 8 | 7 | 5
  Final visit (7 days after the treatment): Normal | 2 | 7 | 3 | 2 | 4
  Final visit (7 days after the treatment): Abnormal not clinically significant | 8 | 3 | 7 | 8 | 6

11. Secondary Outcome: Study Part A: ECGs - PR Interval
Description: PR interval in ms recorded in supine position after 5 min at rest
Time Frame: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  Screening visit: Normal | 3 | 4 | 2 | 3 | 5
  Screening visit: Abnormal, not clinically significant | 7 | 6 | 8 | 7 | 5
  Day 1 (treatment day) at pre-administration: Normal | 1 | 4 | 2 | 2 | 2
  Day 1 (treatment day) at pre-administration: Abnormal, not clinically significant | 9 | 6 | 8 | 8 | 8
  Day 1 (treatment day) at the end of administration: Normal | 2 | 3 | 2 | 2 | 2
  Day 1 (treatment day) at the end of administration: Abnormal, not clinically significant | 8 | 7 | 8 | 8 | 8
  Day 1 (treatment day) at 1 h after the end of administration: Normal | 1 | 2 | 2 | 1 | 2
  Day 1 (treatment day) at 1 h after the end of administration: Abnormal, not clinically significant | 9 | 8 | 8 | 9 | 8
  Day 1 (treatment day) at 2 h after the end of administration: Normal | 0 | 2 | 2 | 2 | 2
  Day 1 (treatment day) at 2 h after the end of administration: Abnormal, not clinically significant | 10 | 8 | 8 | 8 | 8
  Day 1 (treatment day) at 4 h after the end of administration: Normal | 1 | 2 | 1 | 1 | 2
  Day 1 (treatment day) at 4 h after the end of administration: Abnormal, not clinically significant | 9 | 8 | 9 | 9 | 8
  Day 1 (treatment day) at 24 h after the end of administration: Normal | 0 | 4 | 2 | 3 | 5
  Day 1 (treatment day) at 24 h after the end of administration: Abnormal, not clinically significant | 10 | 6 | 8 | 7 | 5
  Final visit (7 days after the treatment): Normal | 2 | 7 | 3 | 2 | 4
  Final visit (7 days after the treatment): Abnormal, not clinically significant | 8 | 3 | 7 | 8 | 6

12. Secondary Outcome: Study Part A: ECGs - RR Interval
Description: RR interval in ms recorded in supine position after 5 min at rest
Time Frame: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  Screening visit: Normal | 3 | 4 | 2 | 3 | 5
  Screening visit: Abnormal, not clinically significant | 7 | 6 | 8 | 7 | 5
  Day 1 (treatment day) at pre-administration: Normal | 1 | 4 | 2 | 2 | 2
  Day 1 (treatment day) at pre-administration: Abnormal, not clinically significant | 9 | 6 | 8 | 8 | 8
  Day 1 (treatment day) at the end of administration: Normal | 2 | 3 | 2 | 2 | 2
  Day 1 (treatment day) at the end of administration: Abnormal, not clinically significant | 8 | 7 | 8 | 8 | 8
  Day 1 (treatment day) at 1 h after the end of administration: Normal | 1 | 2 | 2 | 1 | 2
  Day 1 (treatment day) at 1 h after the end of administration: Abnormal, not clinically significant | 9 | 8 | 8 | 9 | 8
  Day 1 (treatment day) at 2 h after the end of administration: Normal | 0 | 2 | 2 | 2 | 2
  Day 1 (treatment day) at 2 h after the end of administration: Abnormal, not clinically significant | 10 | 8 | 8 | 8 | 8
  Day 1 (treatment day) at 4 h after the end of administration: Normal | 1 | 2 | 1 | 1 | 2
  Day 1 (treatment day) at 4 h after the end of administration: Abnormal, not clinically significant | 9 | 8 | 9 | 9 | 8
  Day 1 (treatment day) at 24 h after the end of administration: Normal | 0 | 4 | 2 | 3 | 5
  Day 1 (treatment day) at 24 h after the end of administration: Abnormal, not clinically significant | 10 | 6 | 8 | 7 | 5
  Final visit (7 days after the treatment): Normal | 2 | 7 | 3 | 2 | 4
  Final visit (7 days after the treatment): Abnormal, not clinically significant | 8 | 3 | 7 | 8 | 6

13. Secondary Outcome: Study Part A: ECGs - QRS Duration
Description: QRS duration in ms recorded in supine position after 5 min at rest
Time Frame: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  Screening visit: Normal | 3 | 4 | 2 | 3 | 5
  Screening visit: Abnormal not clinically significant | 7 | 6 | 8 | 7 | 5
  Day 1 (treatment day) at pre-administration: Normal | 1 | 4 | 2 | 2 | 2
  Day 1 (treatment day) at pre-administration: Abnormal not clinically significant | 9 | 6 | 8 | 8 | 8
  Day 1 (treatment day) at the end of administration: Normal | 2 | 3 | 2 | 2 | 2
  Day 1 (treatment day) at the end of administration: Abnormal not clinically significant | 8 | 7 | 8 | 8 | 8
  Day 1 (treatment day) at 1 h after the end of administration: Normal | 1 | 2 | 2 | 1 | 2
  Day 1 (treatment day) at 1 h after the end of administration: Abnormal not clinically significant | 9 | 8 | 8 | 9 | 8
  Day 1 (treatment day) at 2 h after the end of administration: Normal | 0 | 2 | 2 | 2 | 2
  Day 1 (treatment day) at 2 h after the end of administration: Abnormal not clinically significant | 10 | 8 | 8 | 8 | 8
  Day 1 (treatment day) at 4 h after the end of administration: Normal | 1 | 2 | 1 | 1 | 2
  Day 1 (treatment day) at 4 h after the end of administration: Abnormal not clinically significant | 9 | 8 | 9 | 9 | 8
  Day 1 (treatment day) at 24 h after the end of administration: Normal | 0 | 4 | 2 | 3 | 5
  Day 1 (treatment day) at 24 h after the end of administration: Abnormal not clinically significant | 10 | 6 | 8 | 7 | 5
  Final visit (7 days after the treatment): Normal | 2 | 7 | 3 | 2 | 4
  Final visit (7 days after the treatment): Abnormal not clinically significant | 8 | 3 | 7 | 8 | 6

14. Secondary Outcome: Study Part A: ECGs - QT Interval
Description: QT interval in ms recorded in supine position after 5 min at rest
Time Frame: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  Screening visit: Normal | 3 | 4 | 2 | 3 | 5
  Screening visit: Abnormal, not clinically significant | 7 | 6 | 8 | 7 | 5
  Day 1 (treatment day) at pre-administration: Normal | 1 | 4 | 2 | 2 | 2
  Day 1 (treatment day) at pre-administration: Abnormal, not clinically significant | 9 | 6 | 8 | 8 | 8
  Day 1 (treatment day) at the end of administration: Normal | 2 | 3 | 2 | 2 | 2
  Day 1 (treatment day) at the end of administration: Abnormal, not clinically significant | 8 | 7 | 8 | 8 | 8
  Day 1 (treatment day) at 1 h after the end of administration: Normal | 1 | 2 | 2 | 1 | 2
  Day 1 (treatment day) at 1 h after the end of administration: Abnormal, not clinically significant | 9 | 8 | 8 | 9 | 8
  Day 1 (treatment day) at 2 h after the end of administration: Normal | 0 | 2 | 2 | 2 | 2
  Day 1 (treatment day) at 2 h after the end of administration: Abnormal, not clinically significant | 10 | 8 | 8 | 8 | 8
  Day 1 (treatment day) at 4 h after the end of administration: Normal | 1 | 2 | 1 | 1 | 2
  Day 1 (treatment day) at 4 h after the end of administration: Abnormal, not clinically significant | 9 | 8 | 9 | 9 | 8
  Day 1 (treatment day) at 24 h after the end of administration: Normal | 0 | 4 | 2 | 3 | 5
  Day 1 (treatment day) at 24 h after the end of administration: Abnormal, not clinically significant | 10 | 6 | 8 | 7 | 5
  Final visit (7 days after the treatment): Normal | 2 | 7 | 3 | 2 | 4
  Final visit (7 days after the treatment): Abnormal, not clinically significant | 8 | 3 | 7 | 8 | 6

15. Secondary Outcome: Study Part A: ECGs - QTcB Interval
Description: QTcB interval in ms recorded in supine position after 5 min at rest
Time Frame: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  Screening visit: Normal | 3 | 4 | 2 | 3 | 5
  Screening visit: Abnormal not clinically significant | 7 | 6 | 8 | 7 | 5
  Day 1 (treatment day) at pre-administration: Normal | 1 | 4 | 2 | 2 | 2
  Day 1 (treatment day) at pre-administration: Abnormal not clinically significant | 9 | 6 | 8 | 8 | 8
  Day 1 (treatment day) at the end of administration: Normal | 2 | 3 | 2 | 2 | 2
  Day 1 (treatment day) at the end of administration: Abnormal not clinically significant | 8 | 7 | 8 | 8 | 8
  Day 1 (treatment day) at 1 h after the end of administration: Normal | 1 | 2 | 2 | 1 | 2
  Day 1 (treatment day) at 1 h after the end of administration: Abnormal not clinically significant | 9 | 8 | 8 | 9 | 8
  Day 1 (treatment day) at 2 h after the end of administration: Normal | 0 | 2 | 2 | 2 | 2
  Day 1 (treatment day) at 2 h after the end of administration: Abnormal not clinically significant | 10 | 8 | 8 | 8 | 8
  Day 1 (treatment day) at 4 h after the end of administration: Normal | 1 | 2 | 1 | 1 | 2
  Day 1 (treatment day) at 4 h after the end of administration: Abnormal not clinically significant | 9 | 8 | 9 | 9 | 8
  Day 1 (treatment day) at 24 h after the end of administration: Normal | 0 | 4 | 2 | 3 | 5
  Day 1 (treatment day) at 24 h after the end of administration: Abnormal not clinically significant | 10 | 6 | 8 | 7 | 5
  Final visit (7 days after the treatment): Normal | 2 | 7 | 3 | 2 | 4
  Final visit (7 days after the treatment): Abnormal not clinically significant | 8 | 3 | 7 | 8 | 6

16. Secondary Outcome: Study Part A: ECGs - QTcF Interval
Description: QTcF interval in ms recorded in supine position after 5 min at rest
Time Frame: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  Screening visit: Normal | 3 | 4 | 2 | 3 | 5
  Screening visit: Abnormal not clinically significant | 7 | 6 | 8 | 7 | 5
  Day 1 (treatment day) at pre-administration: Normal | 1 | 4 | 2 | 2 | 2
  Day 1 (treatment day) at pre-administration: Abnormal not clinically significant | 9 | 6 | 8 | 8 | 8
  Day 1 (treatment day) at the end of administration: Normal | 2 | 3 | 2 | 2 | 2
  Day 1 (treatment day) at the end of administration: Abnormal not clinically significant | 8 | 7 | 8 | 8 | 8
  Day 1 (treatment day) at 1 h after the end of administration: Normal | 1 | 2 | 2 | 1 | 2
  Day 1 (treatment day) at 1 h after the end of administration: Abnormal not clinically significant | 9 | 8 | 8 | 9 | 8
  Day 1 (treatment day) at 2 h after the end of administration: Normal | 0 | 2 | 2 | 2 | 2
  Day 1 (treatment day) at 2 h after the end of administration: Abnormal not clinically significant | 10 | 8 | 8 | 8 | 8
  Day 1 (treatment day) at 4 h after the end of administration: Normal | 1 | 2 | 1 | 1 | 2
  Day 1 (treatment day) at 4 h after the end of administration: Abnormal not clinically significant | 9 | 8 | 9 | 9 | 8
  Day 1 (treatment day) at 24 h after the end of administration: Normal | 0 | 4 | 2 | 3 | 5
  Day 1 (treatment day) at 24 h after the end of administration: Abnormal not clinically significant | 10 | 6 | 8 | 7 | 5
  Final visit (7 days after the treatment): Normal | 2 | 7 | 3 | 2 | 4
  Final visit (7 days after the treatment): Abnormal not clinically significant | 8 | 3 | 7 | 8 | 6

17. Secondary Outcome: Study Part A: Clinical Laboratory Tests (Blood Chemistry, Haematology, Urinalysis)
Description: Leukocytes and leukocyte differential count, erythrocytes, haemoglobin, haematocrit, MCV, MCH, MCHC, thrombocytes, electrolytes (sodium, potassium, calcium, chloride, inorganic phosphorus), enzymes (alkaline phosphatase, γ-GT, AST, ALT), substrates/metabolites (total bilirubin, creatinine, glucose, urea, uric acid, total cholesterol, triglycerides), total proteins, urine chemical analysis (pH, specific weight, appearance, color, nitrites, proteins, glucose, urobilinogen, bilirubin, ketones, hematic pigments, leukocytes), urine sediment (analysis performed only if positive: leukocytes, erythrocytes, flat cells, round cells, crystals, cylinders, mucus, bacteria, glomerular erythrocytes). Any abnormalities are recorded.
Time Frame: Screening visit (day of informed consent signature)/final visit (7 days after the treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  Screening visit - blood: Normal | 5 | 2 | 2 | 3 | 1
  Screening visit - blood: Abnormal not clinically significant | 5 | 8 | 8 | 7 | 9
  Screening visit - blood: Abnormal clinically significant | 0 | 0 | 0 | 0 | 0
  Screening visit - urine: Normal | 3 | 3 | 4 | 3 | 2
  Screening visit - urine: Abnormal not clinically significant | 7 | 7 | 6 | 7 | 8
  Screening visit - urine: Abnormal clinically significant | 0 | 0 | 0 | 0 | 0
  Final visit (7 days after the treatment) - blood: Normal | 2 | 4 | 1 | 1 | 0
  Final visit (7 days after the treatment) - blood: Abnormal not clinically significant | 8 | 6 | 8 | 9 | 10
  Final visit (7 days after the treatment) - blood: Abnormal clinically significant | 0 | 0 | 1 | 0 | 0
  Final visit (7 days after the treatment) - urine: Normal | 3 | 3 | 3 | 4 | 3
  Final visit (7 days after the treatment) - urine: Abnormal not clinically significant | 7 | 7 | 7 | 6 | 7
  Final visit (7 days after the treatment) - urine: Abnormal clinically significant | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Study Part A: Cmax
Description: Maximum plasma concentration measured for plasma fosnetupitant, netupitant and its main metabolites (M1, M2 and M3)
Time Frame: Day 1 (treatment day) at pre-administration, at 2, 5, 10, 15, 20, 30 and 45 min and at 1, 1.5, 2, 3, 4, 8, 12, 24 h after the administration
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
ng/mL
  Fosnetupitant | 8486.000 (2095.382) | 8920.000 (1722.892) | 23650.000 (20971.899) | 32540.000 (6607.437) | 37500.000 (11243.270)
  Netupitant | 767.400 (136.572) | 893.400 (283.232) | 1050.100 (260.591) | 1170.700 (276.310) | 1382.700 (315.816)
  Metabolite M1 | 23.910 (5.324) | 22.380 (8.433) | 22.012 (6.687) | 21.930 (6.958) | 22.910 (7.610)
  Metabolite M2 | 135.730 (58.257) | 150.110 (72.607) | 102.450 (44.216) | 118.160 (49.015) | 146.490 (88.541)
  Metabolite M3 | 46.880 (11.936) | 48.450 (17.019) | 46.570 (16.137) | 47.680 (14.446) | 52.100 (27.347)

19. Secondary Outcome: Study Part A: C0
Description: Plasma concentration at the end of the administration measured for plasma fosnetupitant, netupitant and its main metabolites (M1, M2 and M3)
Time Frame: as for outcome 18
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
ng/mL
  Fosnetupitant | 8486.000 (2095.382) | 8920.000 (1722.892) | 23650.000 (20971.899) | 32540.000 (6607.437) | 33557.000 (15972.519)
  Netupitant | 743.100 (173.921) | 893.400 (283.232) | 946.100 (419.234) | 1019.400 (319.820) | 596.810 (383.903)
  Metabolite M1 | 1.714 (2.229) | 1.753 (1.969) | 0.337 (1.066) | 0.000 (0.000) | 0.000 (0.000)
  Metabolite M2 | 28.150 (10.059) | 49.121 (34.243) | 32.300 (22.563) | 25.680 (11.219) | 12.706 (6.689)
  Metabolite M3 | 6.214 (4.144) | 6.799 (2.989) | 0.727 (1.711) | 0.000 (0.000) | 0.000 (0.000)

20. Secondary Outcome: Study Part A: Tmax
Description: Time to achieve the maximum plasma concentration measured for plasma fosnetupitant, netupitant and its main metabolites (M1, M2 and M3)
Time Frame: as for outcome 18
Measure: Median (Full Range); unit: h
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
h
  Fosnetupitant | 0.5 [0.5 to 0.5] | 0.5 [0.5 to 0.5] | 0.25 [0.25 to 0.3] | 0.08 [0.08 to 0.08] | 0.05 [0.033 to 0.08]
  Netupitant | 0.5 [0.5 to 2] | 0.5 [0.5 to 0.5] | 0.25 [0.25 to 0.33] | 0.125 [0.08 to 0.17] | 0.08 [0.08 to 0.17]
  Metabolite M1 | 12 [2 to 24] | 10 [2 to 24] | 12 [1.5 to 24] | 12 [4 to 24] | 12 [8 to 24]
  Metabolite M2 | 2 [2 to 4] | 2 [1.5 to 3] | 2.5 [0.33 to 3] | 2 [1.5 to 3] | 1.75 [1.5 to 4]
  Metabolite M3 | 24 [12 to 24] | 24 [2 to 24] | 24 [12 to 24] | 24 [12 to 24] | 24 [12 to 24]

21. Secondary Outcome: Study Part A: Clast
Description: Last measurable plasma concentration measured for plasma fosnetupitant, netupitant and its main metabolites (M1, M2 and M3)
Time Frame: as for outcome 18
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
ng/mL
  Fosnetupitant | 79.780 (71.819) | 49.410 (35.149) | 97.140 (122.226) | 45.620 (28.083) | 34.330 (16.176)
  Netupitant | 149.150 (111.842) | 122.490 (40.233) | 136.340 (39.724) | 123.740 (28.843) | 137.270 (66.827)
  Metabolite M1 | 21.150 (3.876) | 20.380 (7.875) | 20.532 (6.667) | 19.990 (5.977) | 21.440 (7.826)
  Metabolite M2 | 20.090 (10.519) | 18.850 (7.890) | 14.534 (4.789) | 18.770 (5.515) | 17.067 (7.953)
  Metabolite M3 | 46.370 (12.315) | 48.020 (17.273) | 44.960 (15.634) | 47.080 (14.763) | 52.060 (27.374)

22. Secondary Outcome: Study Part A: Tlast
Description: Time of last measurable plasma concentration measured for plasma fosnetupitant, netupitant and its main metabolites (M1, M2 and M3)
Time Frame: as for outcome 18
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
h
  Fosnetupitant | 0.83 (0.118) | 0.95 (0.23) | 1.075 (1.048) | 0.6 (0.316) | 0.633 (0.35)
  Netupitant | 24 (0) | 24 (0) | 24 (0) | 24 (0) | 24 (0)
  Metabolite M1 | 24 (0) | 24 (0) | 24 (0) | 24 (0) | 24 (0)
  Metabolite M2 | 24 (0) | 24 (0) | 24 (0) | 24 (0) | 24 (0)
  Metabolite M3 | 24 (0) | 24 (0) | 24 (0) | 24 (0) | 24 (0)

23. Secondary Outcome: Study Part A: AUC0-t
Description: Area under the concentration-time curve from time zero to time of last measurable plasma concentration measured for plasma fosnetupitant, netupitant and its main metabolites (M1, M2 and M3)
Time Frame: as for outcome 18
Measure: Mean (Standard Deviation); unit: h x ng/mL
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
h x ng/mL
  Fosnetupitant | 3217.286 (780.235) | 3374.275 (658.088) | 4807.383 (4537.620) | 3662.088 (630.455) | 3839.681 (859.368)
  Netupitant | 5404.315 (1227.399) | 5232.178 (1119.310) | 5792.056 (1520.649) | 5344.307 (1385.625) | 5656.305 (1998.286)
  Metabolite M1 | 468.997 (113.819) | 456.214 (173.046) | 436.089 (142.089) | 426.440 (122.749) | 447.497 (143.611)
  Metabolite M2 | 1234.204 (767.496) | 1260.320 (477.244) | 959.756 (382.755) | 1137.332 (331.659) | 1182.642 (560.829)
  Metabolite M3 | 833.606 (164.142) | 895.624 (304.534) | 831.375 (306.679) | 826.377 (156.114) | 935.410 (441.878)

24. Secondary Outcome: Study Part A: AUC0-24
Description: Area under the plasma concentration-time curve from time zero to 24 h after the administration measured for plasma fosnetupitant, netupitant and its main metabolites (M1, M2 and M3)
Time Frame: as for outcome 18
Measure: Mean (Standard Deviation); unit: h x ng/mL
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
h x ng/mL
  Fosnetupitant | 3228.246 (781.172) | 3382.473 (657.505) | 4833.636 (4577.777) | 3668.069 (631.004) | 3844.251 (859.498)
  Netupitant | 5404.315 (1227.399) | 5232.178 (1119.310) | 5792.056 (1520.649) | 5344.307 (1385.625) | 5656.305 (1998.286)
  Metabolite M1 | 468.997 (113.819) | 456.214 (173.046) | 436.089 (142.089) | 426.440 (122.749) | 447.497 (143.611)
  Metabolite M2 | 1234.204 (767.496) | 1260.320 (477.244) | 959.756 (382.755) | 1137.332 (331.659) | 1182.642 (560.829)
  Metabolite M3 | 833.606 (164.142) | 895.624 (304.534) | 831.375 (306.679) | 826.377 (156.114) | 935.410 (441.878)

25. Secondary Outcome: Study Part A: Terminal Elimination Rate Constant
Description: Terminal elimination rate constant, calculated, if feasible, by log-linear regression using at least 3 points, C0 and Cmax excluded and measured for plasma fosnetupitant, netupitant and its main metabolites (M1, M2 and M3). Calculation was not feasible for M1 and M3, therefore these analytes are not reported in the Outcome Measure Data Table.
Time Frame: as for outcome 18
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
1/h
  Fosnetupitant | 12.157 (0.662) | 11.734 (0.754) | 14.979 (5.582) | 18.613 (3.868) | 19.141 (5.429)
  Netupitant | 0.034 (0.012) | 0.034 (0.007) | 0.033 (0.012) | 0.039 (0.005) | 0.032 (0.014)
  Metabolite M2 | 0.063 (0.014) | 0.061 (0.018) | 0.058 (0.017) | 0.059 (0.013) | 0.061 (0.015)

26. Secondary Outcome: Study Part A: t1/2
Description: Apparent terminal half-life calculated, if feasible, by as ln2/terminal elimination rate constant and measured for plasma fosnetupitant, netupitant and its main metabolites (M1, M2 and M3). Calculation was not feasible for M1 and M3, therefore these analytes are not reported in the Outcome Measure Data Table.
Time Frame: as for outcome 18
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
h
  Fosnetupitant | 0.057 (0.003) | 0.059 (0.004) | 0.080 (0.115) | 0.039 (0.011) | 0.040 (0.017)
  Netupitant | 22.104 (7.005) | 21.356 (4.151) | 25.176 (14.727) | 18.017 (2.747) | 30.061 (24.561)
  Metabolite M2 | 11.538 (2.490) | 12.855 (5.985) | 12.918 (4.023) | 12.468 (3.215) | 12.248 (3.863)

27. Secondary Outcome: Study Part A: Systemic Clearance
Description: Systemic clearance measured for plasma fosnetupitant, netupitant and its main metabolites (M1, M2 and M3). Calculation was not feasible for M1 and M3, therefore these analytes are not reported in the Outcome Measure Data Table.
Time Frame: as for outcome 18
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
mL/h
  Fosnetupitant | 61821.940 (16436.343) | 66942.974 (12370.822) | 65171.229 (21219.721) | 65651.064 (9975.506) | 63748.966 (13353.411)
  Netupitant | 27219.010 (3356.654) | 28693.446 (7660.440) | 24200.268 (6832.625) | 27596.213 (6404.903) | 26994.542 (10531.874)
  Metabolite M2 | 172324.405 (50962.753) | 162039.804 (57537.646) | 211825.621 (68310.261) | 174034.336 (64374.511) | 182468.624 (68658.409)

28. Secondary Outcome: Study Part A: Vz
Description: Apparent volume of distribution in the post-distribution phase measured for plasma fosnetupitant, netupitant and its main metabolites (M1, M2 and M3). Calculation was not feasible for M1 and M3, therefore these analytes are not reported in the Outcome Measure Data Table.
Time Frame: as for outcome 18
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
mL
  Fosnetupitant | 5129.653 (1631.449) | 5765.916 (1352.379) | 4796.595 (1491.027) | 3728.124 (1263.039) | 3572.355 (1199.382)
  Netupitant | 848022.360 (215723.734) | 872978.816 (264673.002) | 772482.708 (205893.262) | 719627.108 (219903.292) | 944544.565 (311425.672)
  Metabolite M2 | 2895427.080 (954908.605) | 2820832.784 (1000428.130) | 4109459.426 (2374558.032) | 3083100.830 (1154481.625) | 3122087.067 (1170365.896)

29. Secondary Outcome: Study Part A: MRT
Description: Mean residence time measured for plasma fosnetupitant, netupitant and its main metabolites (M1, M2 and M3). Calculation was not feasible for M1 and M3, therefore these analytes are not reported in the Outcome Measure Data Table.
Time Frame: as for outcome 18
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
h
  Fosnetupitant | 0.253 (0.001) | 0.254 (0.002) | 0.275 (0.038) | 0.109 (0.014) | 0.086 (0.014)
  Netupitant | 28.529 (9.761) | 26.760 (5.780) | 33.752 (21.148) | 24.493 (3.866) | 40.753 (34.769)
  Metabolite M2 | 14.343 (2.220) | 15.895 (7.651) | 16.347 (5.492) | 16.299 (3.936) | 14.975 (4.858)

ADVERSE EVENTS:
Time Frame: The reporting period for adverse events is the period starting from the time of informed consent signature and lasting until the final visit. Adverse events were collected for each participant for the whole period of the study (i.e., a maximum of 28 days).
Arm/Group | Study Part A - Cohort 1 - Akynzeo | Study Part A - Cohort 1 - Fosnetupitant | Study Part A - Cohort 2 | Study Part A - Cohort 3 | Study Part A - Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 5/10 | 3/10 | 2/10 | 1/10 | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Part A - Cohort 1 - Akynzeo (N=10) | Study Part A - Cohort 1 - Fosnetupitant (N=10) | Study Part A - Cohort 2 (N=10) | Study Part A - Cohort 3 (N=10) | Study Part A - Cohort 4 (N=10)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AST increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
M1 and M3 metabolites on average showed an extent of exposure (AUC) lower than the other analytes. In particular, both metabolites had a significantly longer elimination phase. Indeed, the concentrations of both metabolites were still at a plateau at the end of the sampling period and their elimination kinetics could not be characterized in the present study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-05-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT06840769/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT06840769/SAP_001.pdf